CLINICAL TRIAL: NCT01558843
Title: Sodium Management in Patients With Acute Neurological Injury
Brief Title: Sodium Management in Acute Neurological Injury
Acronym: SANI
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Theresa Human-Murphy, Pharm.D., BCPS, Washington University School of Medicine
Other Study IDs: 201203034
Record Dates: First submitted 2012-03-17; First posted 2012-03-20 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: This Study is to Understand the Current Practice of Sodium Management in Acute Neurological Injury
Keywords: Sodium Management; Neurointensive Care; Hyponatremia
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- traumatic brain injury
- aneurysmal subarachnoid hemorrhage
- intracerebral hematoma
- brain tumor

SUMMARY:
This multicenter, observational, study will enroll severe neurologically injured patients both prospectively and retrospectively. The aims are to identify the percent of neurocritical care patients with sodium levels ≤ 135 mEq/L, describe treatment strategies employed, determine the correlation of clinical factors (i.e. GCS, ICP) with serum sodium concentrations in patients prior to sodium altering therapy, and evaluate outcomes through evaluation of length of stay, discharge disposition, and modified Rankin score (mRS).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years of age
* admitted to an intensive care unit for more than 48 hours
* ICD-9 codes for aneurysmal SAH, TBI, IPH, or intracranial tumor.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients identified for enrollment will be age ≥ 18 years of age, admitted to an intensive care unit for more than 48 hours with ICD-9 codes for aneurysmal SAH, TBI, IPH, or intracranial tumor.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2016-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Brophy, Pharm.D, Principal Investigator — VCU; Theresa Murphy-Human, Pharm.D., Principal Investigator — Washington University School of Medicine
Locations (17):
- United States (17):
  - Hartford Hospital, Hartford, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Jackson Memorial Hospital, Miami, Florida
  - Memorial University Medical Center, Savannah, Georgia
  - University of Chicago, Chicago, Illinois
  - Via Christi Hospital, Wichita, Kansas
  - UK Healthcare, Lexington, Kentucky
  - The Johns Hopkins hospital, Baltimore, Maryland
  - Detroit Receiving Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - St Louis University Hospital, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - UC Health -University Hospital, Cincinnati, Ohio
  - University of Tennessee, Knoxville, Tennessee
  - University of Virginial Health System, Charlottesville, Virginia
  - Virginial Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided